CLINICAL TRIAL: NCT02186639
Title: Exhaled Breath Analysis in Patients With COPD by Secondary Electrospray Ionization - Mass Spectrometry (SESI-MS)
Brief Title: Breath Analysis in Chronic Obstructive Lung Disease (COPD)
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Collaborators: Swiss National Science Foundation (Other)
Responsible Party: Sponsor
Other Study IDs: KEK-ZH-Nr. 2014-0088
Record Dates: First submitted 2014-07-02; First posted 2014-07-10 (Estimated); Last update posted 2018-03-29 (Actual); Status verified 2018-03

CONDITIONS: COPD
Keywords: exhaled breath; volatile organic compounds (VOCs); SESI-MS
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- COPD: 40 COPD patients (20 non-frequent and 20 frequent-exacerbators). No intervention.
- Controls: Subjects with no apparent lung disease and normal lung function testing. Matched for age, gender and smoking history (pack years).
  No intervention.

SUMMARY:
To answer the question whether a disease specific profile of breath in patients with COPD can be detected by an untargeted metabolomic study using exhaled breath analysis by mass spectrometry.

DETAILED DESCRIPTION:
This is an observational study comparing the volatile organic compounds (VOCs) in exhaled breath between COPD patients and matched control subjects (age, gender, smoking-state). 40 COPD patients (20 non-frequent, 20 frequent exacerbators) and 40 matched controls will be examined by SESI-MS on the composition of exhaled breath for identification of COPD specific markers.

ELIGIBILITY:
Inclusion Criteria:

* confirmed COPD GOLD stage I-IV, based on a post-bronchodilator spirometry (FEV1/FVC < 0.7) performed within the last 6 months
* age between 18 and 80 years at study entry
* healthy controls: normal spirometry

Exclusion Criteria:

* COPD exacerbation within the last 6 weeks
* any lung disease other than COPD
* acute inflammatory disease (e.g. common cold) within the last 6 weeks
* acute or chronic hepatic disease
* renal failure or renal replacement therapy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients will be recruited in primary, secondary and tertiary care clinics. Healthy controls will be recruited from a community sample.
Sampling Method: Probability Sample
Enrollment: 40 (Actual)
Dates: Start 2014-06; Primary Completion 2016-12 (Actual); Study Completion 2017-11 (Actual)

PRIMARY OUTCOMES:
COPD-specific mass spectrometric exhaled breath pattern | baseline

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm Kohler, Prof., Principal Investigator — University Hospital Zurich, Pulmonary Division
Locations (1):
- University Hospital Zurich, Pulmonary Division, Zurich, Switzerland

REFERENCES:
- [Derived] Gaugg MT, Nussbaumer-Ochsner Y, Bregy L, Engler A, Stebler N, Gaisl T, Bruderer T, Nowak N, Sinues P, Zenobi R, Kohler M. Real-Time Breath Analysis Reveals Specific Metabolic Signatures of COPD Exacerbations. Chest. 2019 Aug;156(2):269-276. doi: 10.1016/j.chest.2018.12.023. Epub 2019 Jan 24. PMID 30685334